CLINICAL TRIAL: NCT02987361
Title: Effects of Transcranial Direct Current Stimulation on Hemiplegic Upper Extremity Function After Strokes
Brief Title: Effect of tDCS on Upper Extremity After Strokes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Myoung Hwan Ko, Professor, Chonbuk National University Hospital
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: CBNUH_MDCTC_2015_tDCS
Record Dates: First submitted 2016-08-31; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- treatment group 1 (Experimental): anodal stimulation on the lesioned primary motor cortex DC-STIMULATOR PLUS
  Interventions: Device: DC-STIMULATOR PLUS
- treatment group 2 (Experimental): cathodal stimulation on the non-lesioned primary motor cortex DC-STIMULATOR PLUS
  Interventions: Device: DC-STIMULATOR PLUS
- treatment group 3 (Experimental): dual stimulation such as anodal stimulation on the lesioned side and cathodal stimulation on the non-lesioned side DC-STIMULATOR PLUS
  Interventions: Device: DC-STIMULATOR PLUS
- sham group (Sham Comparator): sham group
  Interventions: Device: DC-STIMULATOR PLUS

INTERVENTIONS:
Device: DC-STIMULATOR PLUS — 2mA for 20minutes a day, 5 days per weeks, totally 2 weeks
  Other Names: tDCS

SUMMARY:
The investigators hypothesize that transcranial direct current stimulation (tDCS) can improve upper limb motor recovery in the sub-acute phase of stroke patients.

This is a randomized, controlled, double blind, cross-over, multicentre, clinical trial.

DETAILED DESCRIPTION:
The investigators hypothesize that transcranial direct current stimulation (tDCS) can improve upper limb motor recovery in the sub-acute phase of stroke patients.

This is a randomized, controlled, double blind, cross-over, multicentre, clinical trial.

Informed consent was obtained from all participants and procedures were conducted according to the Declaration of Helsinki. The protocol was approved by the Chonbuk National Uni. Hospital IRB, KOREA.

Seventy-two stroke patients in the sub-acute phase will be recruited in three centers of neurorehabilitation in republic of Korea.

Patients will be randomly divided to four groups; group1 is anodal stimulation on the lesioned primary motor cortex, group 2 is cathodal stimulation on the non-lesioned primary motor cortex, group 3 is dual stimulation such as anodal stimulation on the lesioned side and cathod stimulation on the non-lesioned side, and group 4 is shame stimulation group.

The stimulation will be conducted 2mA for 20 minute a day, 5 days per weeks, totally 2 weeks.

Fugl-Meyer upper motor score will be measured as a primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-85
2. Unilateral Stroke patients
3. Inclusion must be in the sub-acute phase defined as within 48hr-4 weeks after stroke
4. Patients who have evoked motor potentials on the first dorsal interossei muscles on hemiplegic hand
5. The patient has subscribed the informed consent

Exclusion Criteria:

1. Insert a metal object on the head
2. Convulsive disorders
3. History of brain diseases other than stroke

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Motor Score change | before treatment, 48 hours after treatment, 4 weeks after treatment

SECONDARY OUTCOMES:
Manual Muscle Test (MMT) change | before treatment, 48 hours after treatment, 4 weeks after treatment
Range of Motion (ROM) change | before treatment, 48 hours after treatment, 4 weeks after treatment
Korean version Modified Bathel Index (KMBI) change | before treatment, 48 hours after treatment, 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Myoung Hwan Ko, MD, PhD, Principal Investigator — 634-18, Geumam-dong, Deokjin-gu, Jeonju, Jeonbuk, 561-712 Republic of Korea
Locations (1):
- Kim Yeon Hee, Seoul, Ilwon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided